CLINICAL TRIAL: NCT01204216
Title: Does Variation in Mean Red Cell Age Impact HbA1C Interpretation?
Brief Title: Effect of Red Blood Cell Survival on a Commonly Used Diabetes Lab Test-HbA1c
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: technical barriers to completing the original design within the funding period
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDA-006-09S; 09100601 (Other Grant/Funding Number: University of Cincinnati)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Impaired Fasting Glucose; Prediabetes
Keywords: Hemoglobin A1c; HbA1c; glycated serum proteins; fructosamine; glycated albumin; glycation gap
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aim 1 (Active Comparator): Subjects in this arm will be 10 people without diabetes as well as 10 people with diabetes and stable glycemic control. Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  Interventions: Biological: re-infusion of biotin labeled cells
- Aim 2 (Active Comparator): For Aim 2, 10 additional subjects with diabetes in poor glycemic control will be studied initially and then again in improved glycemic control after at least 8 months (with up to 5 additional subjects entered as needed to ensure 10 completed paired studies) to assess the potential role of MRBC variation in the discordances seen between HbA1c and blood glucose testing. Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  Interventions: Biological: Re-infusion of biotin labeled cells; Behavioral: Diabetes education/diabetes medication adjustment

INTERVENTIONS:
Biological: re-infusion of biotin labeled cells — Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  These experiments require a series of small, precisely timed post-infusion blood samples over a period of 4 months, with each subject undergoing the procedure twice separated by an interval of at least 8 month
  Arms: Aim 1
Biological: Re-infusion of biotin labeled cells — Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  These experiments require a series of small, precisely timed post-infusion blood samples over a period of 4 months, with each subject undergoing the procedure twice separated by an interval of at least 8 months.
  small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  Arms: Aim 2
Behavioral: Diabetes education/diabetes medication adjustment — Between the initial 3-4 month trial period and the second infusion of biotin labeled cells approximately 8 months later,subjects will receive diabetes education from a CDE. In addition,if needed, diabetes medications may be adjusted by the study endocrinologist to improve subject's glycemic control.
  Arms: Aim 2

SUMMARY:
Prevention of complications in veterans with diabetes depends heavily on assessment of blood glucose and HbA1c. The HbA1c is a blood test that measures the exposure of hemoglobin (Hb) to a person's average blood glucose over the lifespan of a red blood cell (RBC). The test is heavily relied upon as a measure of blood glucose control. It is normally assumed that all people (those with and without diabetes) have a narrow range of red blood cell survival. It has been recently shown that this is not a valid assumption.

A more precise test of red blood cell survival, using a biotin label method, demonstrated a substantial difference of red blood cell survival among otherwise normal people. There is sufficient difference in red blood cell survival to alter the estimate of glycemic control from the HbA1c test by as much as 30 per cent. This introduces concern that HbA1c values do not mean the same thing in a significant number of people.

Although the evidence is clear that there is variation in RBC survival among people, attributing this variation to differences between individuals depends on answering several simple questions which surprisingly remain unanswered: whether RBC survival is stable over time within an individual and whether blood glucose control affects its stability. Therefore, the goal of the proposed studies is to define these characteristics.

DETAILED DESCRIPTION:
The first Specific Aim tests the hypothesis that mean RBC age is stable in subjects without diabetes and in subjects with diabetes at stable glycemic control. The second Specific Aim tests the hypothesis that mean RBC age will not change in subjects with diabetes studied initially in poor glycemic control, and again after being treated to stable, improved glycemic control for >8 months. To accomplish the two aims, RBC survival and mean blood glucose will be determined at two times separated by at least eight months in 10 subjects without diabetes, 10 subjects with diabetes and stable glycemic control, and up to 15 subjects with diabetes in initial poor glycemic control in order to re-study 10 subjects subsequently in improved glycemic control. The RBC survival will be measured using the same novel biotin RBC label in conjunction with mean glucose determination by continuous glucose monitoring. Mean blood glucose will be assessed using blood glucose testing meter , continuous glucose monitoring equipment, HbA1c, fructosamine and glycated albumin determinations HbA1c is the most highly valued clinical test for long term monitoring of glycemic control and the prediction of diabetes complications risk is relied upon for hundreds of thousands of clinical decisions made every year in veterans with diabetes. The proposed studies, by further defining RBC survival stability necessary to develop a new approach to HbA1c interpretation, therefore has the potential to dramatically support the Department of Veterans Affairs in its mission to reduce the burden of diabetes and its complications

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between ages 18 and 85 for Aim 1 and between 18 and 80 years for Aim 2 and non-pregnant
* Subjects with both types 1 and 2 diabetes
* Subjects without diabetes (as determined by an OGTT test at screening)
* veterans receiving care at VAMC will be given preference but open to both veterans and non-veterans.

Exclusion Criteria:

* known hemoglobinopathy or RBC disorder
* positive pregnancy test (in women of child-bearing potential or are breast feeding or planning pregnancy during the course of the study;
* baseline serum creatinine >1.5 mg/dl
* CBC outside the normal range
* history of GI blood loss or coagulopathy
* urine microalbumin >100 mcg/mg creatinine (spot collection);
* transaminases >3 X the upper limit of normal
* presence of serum antibodies to biotinylated proteins (which could interfere with the biotin RBC labeling protocol)
* greater than or equal to NYHA stage 3 heart failure;
* active infection;
* known rheumatologic disease
* uncontrolled hypo-or hyperthyroidism or an underlying illness known to be associated with either body wasting or changes in serum proteins
* plans to move out of the area within the time frame of the Aim for which they are recruited
* unwillingness to perform self monitoring of blood glucose

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Cohen, MD, Principal Investigator — Cincinnati VA Medical Center, Cincinnati, OH
Locations (1):
- Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Cohen RM, Franco RS, Khera PK, Smith EP, Lindsell CJ, Ciraolo PJ, Palascak MB, Joiner CH. Red cell life span heterogeneity in hematologically normal people is sufficient to alter HbA1c. Blood. 2008 Nov 15;112(10):4284-91. doi: 10.1182/blood-2008-04-154112. Epub 2008 Aug 11. PMID 18694998
- [Background] Cohen RM, Lindsell CJ. When the blood glucose and the HbA(1c) don't match: turning uncertainty into opportunity. Diabetes Care. 2012 Dec;35(12):2421-3. doi: 10.2337/dc12-1479. No abstract available. PMID 23173128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol interrupted due to IND closure, precluding completion of the originally described protocol.
Groups:
- Aim 1: Subjects in this arm will be 10 people without diabetes as well as 10 people with diabetes and stable glycemic control. Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  re-infusion of biotin labeled cells: Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  These experiments require a series of small, precisely timed post-infusion blood samples over a period of 4 months, with each subject undergoing the procedure twice separated by an interval of at least 8 months.
- Aim 2: 10 additional subjects with diabetes in poor glycemic control will be studied initially and then again in improved glycemic control after at least 8 months (with up to 5 additional subjects entered as needed to ensure 10 completed paired studies) to assess the potential role of MRBC variation in the discordances seen between HbA1c and blood glucose testing. Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  Re-infusion of biotin labeled cells: Subjects will participate in experiments involving re-infusion of biotin-labeled cells in which a small volume (< 10 ml) of autologous, biotinylated erythrocytes will be re-infused to determine cell lifespan and in vivo HbA1c formation rate.
  These experiments require a series of small, precisely timed post-infusion blood samples over a period of 4 months, with each subject undergoing the procedure twice separated by an interval of at least 8 months.
  Diabetes education/diabetes medication adjustment: Between the initial 3-4 month trial period and the second infusion of biotin labeled cells approximately 8 months later, subjects will receive diabetes education from a CDE. In addition, if needed, diabetes medications may be adjusted by the study endocrinologist to improve subject's glycemic control.
Period: Overall Study
Arm/Group | Aim 1 | Aim 2
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Protocol interrupted due to IND closure, precluding completion of the originally described protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 1 | Aim 2 | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Specific Aim 1: To Determine the Stability of MRBC (Mean RBC Age)Over Time at Stable Glycemia. The Hypothesis is MRBC Will be Stable in Subjects Without Diabetes and in Subjects With Diabetes at Stable Glycemic Control.
Description: The investigators will determine MRBC and MBG (by both 7 point profile and continuous glucose monitoring), twice in 10 subjects without diabetes and in 10 subjects with diabetes at stable glycemic control. Since the time course study for following the disappearance of re-infused labeled RBCs is approximately 4 months, performing the biotin labeling of the cells for the second study at least 8 months after completion of sampling for the first, effectively samples MRBC at two time points at least one year apart.
Time Frame: Baseline and 8 months later
Population: Protocol interrupted due to IND termination. The data necessary to conduct analysis was not collected.
Arm/Group | Aim 1 | Aim 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Specific Aim 2: To Determine the Impact of Glycemic Control on MRBC.
Description: Up to 15 subjects participating in Aim 2 will be studied initially in poor glycemic control, while their second biotin/glucose monitoring study will be performed at least 8 months later after achieving stable glycemic control. If RBC survival varies, and in particular if it varies with glycemic control, then the relationship between HbA1c and MBG will change. Several studies have reported that HbA1c rises linearly with MBG until there is the appearance of a plateau suggesting a saturation maximum.
Time Frame: Baseline and 8 months later
Population: Protocol interrupted due to IND termination. The data necessary to conduct analysis was not collected.
Arm/Group | Aim 1 | Aim 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events assessed throughout the approximately 4 month duration of study and for 3 months after study completion.
Description: Protocol interrupted due to IND termination. Analysis not conducted.
Arm/Group | Aim 1 | Aim 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

LIMITATIONS AND CAVEATS:
The protocol interrupted due to termination of IND. Insufficient time to complete the protocol within the term despite new IND for same biotin labelling of RBCs. Remaining grant funds applied to similar physiologic studies using 15N-glycine labelling of RBCs. see PMID: 25293624 for results. Those results led to funding of NIH Grant 1R01DK123330-01A1 "Towards optimizing diabetes management and diagnosis by personalizing HbA1c targets."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No